CLINICAL TRIAL: NCT04332367
Title: Phase II, Single-Arm Study Of Carboplatin, Weekly Taxane, And Ramucirumab In Advanced Non-Squamous Non-Small Cell Lung Cancer (NSCLC) After Progressive Disease On Maintenance Pemetrexed And/Or Pembrolizumab
Brief Title: Carboplatin, Taxane And Ramucirumab for Patients With NSCLC After Pemetrexed or Pembrolizumab Maintenance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 05519; IRB833759 (Other: University of Pennsylvania)
Record Dates: First submitted 2020-03-11; First posted 2020-04-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Albumin-Bound Paclitaxel; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carboplatin, Taxane And Ramucirumab (Experimental): Carboplatin AUC 5 IV every 3 wks, Paclitaxel 80 mg/m2 IV days 1 and 8 every 3 weeks, and Ramucirumab 10 mg/kg IV every 3 weeks
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Ramucirumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin IV
  Other Names: Paraplatin
Drug: Paclitaxel — Paclitaxel IV
  Other Names: Abraxane, Taxol
Drug: Ramucirumab — Ramucirumab IV
  Other Names: Cyramza

SUMMARY:
The purpose of this study is to determine if the combination of the three anti-cancer drugs carboplatin, paclitaxel, and ramucirumab is helpful in shrinking tumors or delaying tumor growth in participants with non-small cell lung cancer. This study will also assess whether it is safe to combine these drugs.

ELIGIBILITY:
Inclusion Criteria:

* Advanced non-squamous NSCLC (Stage IV or recurrent after initial curative intent therapy) in adults age 18 or older
* Prior exposure to 4-6 cycles of Pem/Carbo/Pembro and PD after at least 18 weeks of maintenance Pemetrexed, Pembrolizumab or the combination of the two.
* PS 0-1

Exclusion Criteria:

* Presence of a driver mutation that is susceptible to targeted therapy
* Other active invasive malignancy requiring ongoing therapy
* Grade 2 or higher sensory neuropathy
* Evidence of untreated brain metastases
* History of bleeding diatheses or recent, antecedent hemoptysis (> 1/2 teaspoon in prior 2 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To estimate overall response rate | 3 years
  Overall response rate (ORR) as determined by RECIST criteria. Response will be defined by a complete response (CR) or partial response (PRO), confirmed or unconfirmed.

SECONDARY OUTCOMES:
Progression-free survival | From first dose of study drug until progressive disease, death or last assessment contact, whichever comes first, an average of 1-2 years
  Progression-free survival (PFS) defined as the duration from the first study dose of study drug until progressive disease, death or last assessment contact whichever comes first.
Overall Survival | from the first dose of study drug until death, last observation or contact, an average of 1-2 years
  Overall Survival (OS) is defined as the time from the first dose of study drug until death due to any cause or last observation or contact.
Safety Evaluations: number of Grade ≥ 3 as determined by CTCAE v 5.0 | Initiation through 30 days following the last administration of study treatment.
  Toxicity will be estimated by the number of Grade ≥ 3 as determined by CTCAE v 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Melina Marmarelis, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT04332367/ICF_000.pdf